CLINICAL TRIAL: NCT02574741
Title: Augmenting Language Interventions in ASD: A Translational Approach (ACE Project 3)
Brief Title: Combination Treatment for Augmenting Language in Children With ASD
Acronym: PIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, James McCracken, Director/Vice Chair, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-000726
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Behavior Therapy; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aripiprazole (Active Comparator): Aripiprazole oral solution (1mg/mL) for 12 weeks. dosages range from 2-10mg per day.
  Interventions: Behavioral: Behavioral Therapy; Drug: Aripiprazole
- Placebo (Active Comparator): 50% will be randomized to placebo.
  Interventions: Behavioral: Behavioral Therapy; Drug: Placebo
- Behavioral Intervention (Active Comparator): All subjects will receive behavioral therapy, in addition to either active study drug (aripiprazole) or placebo.
  Interventions: Behavioral: Behavioral Therapy; Drug: Aripiprazole; Drug: Placebo

INTERVENTIONS:
Behavioral: Behavioral Therapy — Thrice-weekly individually based language JAE-EMT intervention will be provided by a trained therapist and taught to the child and their caregivers. A total of 36 sessions will be provided over 12 weeks, with 2 per week at UCLA, and one session per week in the home.
  Other Names: language intervention
Drug: Aripiprazole — 50% of the subjects will be randomized to aripiprazole (active study medication)
  Other Names: abilify
  Arms: Aripiprazole; Behavioral Intervention
Drug: Placebo — 50% of the subjects will be randomized to placebo (inactive study medication).
  Other Names: inactive study medication
  Arms: Behavioral Intervention; Placebo

SUMMARY:
The study will consist of two main elements: the enrollment of 72 children aged 6-11 years with ASD and low language competency to receive a thrice-weekly one hour language intervention for 12 weeks; and, beginning at the same time, subjects will be equally randomized to receive either aripiprazole (Abilify) (flexibly dosed from 2-10 mg per day) or placebo for 12 weeks.

DETAILED DESCRIPTION:
Following screening for eligibility and baseline, study visits will be scheduled three times per week, with 2 sessions on-site at UCLA and one at home for parent training (allowing flexibility, as needed); study physician visits will occur once weekly for 6 weeks, then biweekly. Screening procedures may be completed in one or two visits, and measures obtained in other UCLA clinical or research setting may be used if assessments were done within one month of screening. Major outcome assessments will occur at baseline (Week 0), mid-point (Week 6), and final week (Week 12) by study personnel blind to visit number and drug group assignment; minor assessments will occur weekly along with study physician assessments occurring weekly for side effect and compliance checks. EEG will occur at or prior to baseline and at Visit 36 (Wk12). Arrangements will be made to transfer participants to standard clinical care following visit 36. Six months after visit 36, families will be seen for final follow-up assessments of language usage, social communication, overall functioning, health and ongoing treatment.

ELIGIBILITY:
Inclusion criteria:

* boys and girls ages 5-11 years;
* criteria for autistic disorder or PDD-NOS as defined by DSM-IV-TR and confirmed by clinical examination and ADI-R, ADOS;
* low language usage as defined by <30 functional words obtained from a natural language sample, parent report, and standardized tests;
* present placement in a comprehensive educational/intervention setting.

Exclusion criteria:

* any medical condition that would interfere with intervention outcomes during a 12 week study period (eg., active seizures within 3 months);
* genetic disorders such as Fragile X, Down syndrome, or tuberous sclerosis;
* sensory impairments such as deafness or blindness;
* existing or anticipated need for concomitant psychotropic medication (specifically stimulants, atomoxetine) during study participation( allowed medication include: antidepressants, anticonvulsants, guanfacine, clonidine, supplements, melatonin, diphenhydramine);
* severe aggression or self-injurious behavior;
* DQ <18 months as assessed by the Leiter-Revised or Mullen.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2012-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of words as assessed in a naturalistic language assessment | 12 weeks post baseline
  word usage coded as assessed by a clinician-administered assessment

CONTACTS AND LOCATIONS:
Overall Officials: James McCracken, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States